CLINICAL TRIAL: NCT03340454
Title: Patient-Centered Cancer Prevention In Chinese Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-01446; 2U54MD000538 (NIH)
Record Dates: First submitted 2017-11-06; First posted 2017-11-13 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: H. Pylori Infection
Keywords: H. pylori; H. pylori infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health systems-level intervention (Active Comparator): using electronic health record (EHR)-based tools to facilitate H. pylori test-and-treat strategies;
  Interventions: Other: Test-and-treat EHR-CHW intervention
- CHW-led patient navigation program (Active Comparator): a community-engaged culturally and linguistically adapted CHW-led patient navigation program we are currently pilot testing for feasibility and acceptability
  Interventions: Other: Usual care of EHR-only intervention

INTERVENTIONS:
Other: Test-and-treat EHR-CHW intervention — a health systems-level intervention using electronic health record (EHR)-based tools to facilitate H. pylori test-and-treat strategies
  Arms: Health systems-level intervention
Other: Usual care of EHR-only intervention — a community-engaged culturally and linguistically adapted CHW-led patient navigation program we are currently pilot testing for feasibility and acceptability.
  Arms: CHW-led patient navigation program

SUMMARY:
This study will assess the efficacy, adoption, and impact of an integrated intervention to improve adherence to recommended stomach cancer prevention guidelines (H. pylori test-and-treat) for at-risk Chinese Americans in NYC. The integrated multifaceted theory-based intervention involves: 1) a health systems-level intervention using electronic health record (EHR)-based tools to facilitate H. pylori test-and-treat strategies; and 2) a community-engaged culturally and linguistically adapted CHW-led patient navigation program we are currently pilot testing for feasibility and acceptability. Using a 2-arm randomized controlled trial (RCT) design, > 144 Chinese American patients across NYC safety net hospital endoscopy clinics and primary health centers will participate.

ELIGIBILITY:
Inclusion Criteria:

* self identifies as Chinese American
* is an outpatient aged 21 years and older (adult)
* plans to continue to live in the region during the next 12 months;
* is willing to be randomized to either treatment or control groups
* has a confirmed diagnosis of H. pylori infection by at least one of the following methods: C-urea breath test, histology, rapid urease test or bacterial culture, fecal stool antigen test or other clinically approved H. pylori infection diagnostic test.

Exclusion Criteria:

* advanced chronic disease that would not allow the patient to complete follow-up or attend visits;
* allergy to any of the study drugs;
* pregnancy or currently breastfeeding
* taking antibiotics or bismuth salts within 2 weeks before the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simona Kwon, DrPH,MPH, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Systems-level Intervention | CHW-led Patient Navigation Program
Started | 67 | 68
Completed | 67 | 64
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Systems-level Intervention | CHW-led Patient Navigation Program | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Continuous [Mean (Full Range); unit: years] | 44 [23 to 81] | 42 [25 to 69] | 43.5 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 31 | 30 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 67 | 64 | 131
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 67 | 64 | 131
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 67 | 64 | 131

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Eradication of H. Pylori (ITT)
Description: Measured using breath ammonia measurement, fecal stool antigen test or other clinically approved H. pylori infection diagnostic test. Data extracted from patient EHR. Includes positive results for those with self-reported or missing results.
Time Frame: Up to Month 3-Post Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Health Systems-level Intervention | CHW-led Patient Navigation Program
Number analyzed (Participants) | 67 | 64
Participants | 49 | 54

2. Secondary Outcome: Number of Participants With Eradication of H. Pylori (Clinically Confirmed)
Description: Measured using breath ammonia measurement, fecal stool antigen test or other clinically approved H. pylori infection diagnostic test. Data extracted from patient EHR.
Time Frame: Up to Month 3-Post Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Health Systems-level Intervention | CHW-led Patient Navigation Program
Number analyzed (Participants) | 56 | 59
Participants | 49 | 54

3. Secondary Outcome: Change in Ottawa Decision Self-Efficacy Scale Score From Baseline to 6 Months
Description: Participants completed the Ottawa Decision Self-Efficacy Scale, which assessed participants' confidence in making an informed choice, at baseline and 6-month follow-up. The scale consists of 11 questions on a 5-point Likert scale from 0 (not at all confident) to 4 (very confident). The raw score is the sum of responses. The raw score is converted to a standardized total score that ranges from 0 to 100; higher total scores indicate greater decision self-efficacy.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Systems-level Intervention | CHW-led Patient Navigation Program
Number analyzed (Participants) | 60 | 57
score on a scale | 5 (13.59) | 5.7 (11.77)

4. Secondary Outcome: Change in Medication Adherence Report Scale (MARS-5) Score From Baseline to Month 6
Description: Participants completed the MARS-5 self-assessment of medication adherence at baseline and 6-month follow-up. One item assessed unintentional non-adherence, while four items assessed intentional non-adherence. Participants indicated how often each statement applied to them in the past month on a 5-point Likert scale (1=always, 2=often, 3=sometimes, 4=rarely, 5=never), resulting in a total score ranging from 5 to 25. Adherence is defined as a score of 25.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Systems-level Intervention | CHW-led Patient Navigation Program
Number analyzed (Participants) | 62 | 57
score on a scale | 0.58 (2.69) | 0.77 (2.95)

5. Secondary Outcome: Change in Stomach Cancer Knowledge Between Baseline and 6-months
Description: Participants were asked about associations with the risk of getting stomach cancer (alcohol, spicy food, stress, family history, h. pylori infection, smoking, salty food, being physically inactive, pickled food, food high in sugar). True or false was chosen. Variables were recoded to correct (1) and incorrect (0), and summed for a final score (0-10, 10=highest knowledge)
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Systems-level Intervention | CHW-led Patient Navigation Program
Number analyzed (Participants) | 60 | 57
score on a scale | 1.58 (2.25) | 3.25 (2.9)

6. Secondary Outcome: Change in H. Pylori Knowledge Between Baseline and 6-months
Description: Participants were asked about associations with h. pylori (blood, untreated/contaminated water, rats, mosquitoes, contaminated food, vomit, poor sanitation). True or false was chosen. Variables were recoded to correct (1) and incorrect (0), and summed for a final score (0-7, 7=highest knowledge)
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Systems-level Intervention | CHW-led Patient Navigation Program
Number analyzed (Participants) | 61 | 59
score on a scale | 1.03 (2) | 2.56 (2.5)

7. Secondary Outcome: Change in PROMIS Global Physical Health T-Score Between Baseline and 6-months
Description: Participants completed the PROMIS Global Physical Health Scale, which assessed participants' physical health, at baseline and 6-month follow-up. Four questions assessed global physical health. Three questions were administered using five-category response scales, and one item used a response scale of 0-10 that was recoded to five categories. Responses are recoded into t-scores, which rescales the raw sum score into a standardized score from 0-100, with a mean of 50 and a standard deviation of 10. Higher scores indicate more of the concept being measured.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Health Systems-level Intervention | CHW-led Patient Navigation Program
Number analyzed (Participants) | 61 | 58
T-score | -1.1 (2.71) | 1.27 (8.27)

8. Secondary Outcome: Change in PROMIS Global Mental Health T-Score Between Baseline and 6-months
Description: Participants completed the PROMIS Global Mental Health Scale, which assessed participants' mental health, at baseline and 6-month follow-up. Four questions assessed global mental health, and all were administered using five-category response scales. Responses are recoded into t-scores, which rescales the raw sum score into a standardized score from 0-100, with a mean of 50 and a standard deviation of 10. Higher scores indicate more of the concept being measured.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Health Systems-level Intervention | CHW-led Patient Navigation Program
Number analyzed (Participants) | 61 | 57
T-score | 0.69 (6.84) | 3.13 (6.07)

ADVERSE EVENTS:
Time Frame: 6 Months
Description: Systematic assessment through standard questionnaire
Arm/Group | Health Systems-level Intervention | CHW-led Patient Navigation Program
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/68
Other Adverse Events (participants affected / at risk) | 0/67 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT03340454/Prot_SAP_000.pdf